CLINICAL TRIAL: NCT07118917
Title: Does a Prior COVID-19 Infection Affect Lung Dynamics During Thoracic Anesthesia?
Brief Title: COVID-19 Infection and Thoracic Anesthesia?
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Professor, Ankara University
Other Study IDs: 2024/667
Record Dates: First submitted 2025-06-24; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-06

CONDITIONS: COVID - 19; Thoracic Anesthesia; Mechanical Power
MeSH Terms: conditions — COVID-19 | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive: COVID-19 positive patients
  Interventions: Other: Prehabilitation
- COVID-19 negative: COVID-19 negative
  Interventions: Other: No postponement

INTERVENTIONS:
Other: Prehabilitation — Patients with COVID-19 history postponed for the surgery according to multidisciplinary decision.
  Groups: COVID-19 positive
Other: No postponement — Patients who were COVID negative proceeded for surgery
  Groups: COVID-19 negative

SUMMARY:
SARS-CoV-2 has infected more than 776 million people worldwide, raising concerns about its impact on patients with lung cancer, the most common cancer in men and the second most common cancer in women. Previous studies have suggested that COVID-19 may worsen lung dysfunction in patients undergoing surgery and that the coexistence of COVID-19 and lung cancer increases the risk of complications and mortality. It has been recommended that surgery be delayed after COVID-19 infection to reduce postoperative risk. This study examined the effects of prior COVID-19 infection on respiratory mechanics in patients undergoing thoracic surgery for lung cancer.

DETAILED DESCRIPTION:
COVID-19 positivity was confirmed in 53 patients via SARS-CoV-2 RT-Prowhite, and the remaining 57 patients were classified as COVID-19 negative on the basis of a lack of prior positive PCR tests and the absence of COVID-19 symptoms in medical records. Statistical analysis was performed via SPSS Statistics for Windows, Version 17.0 (Chicago: SPSS Inc.). The Shapiro-Wilk test was used to assess the normality of the data distribution, a standard approach to determine the appropriateness of parametric versus nonparametric tests. For variables that did not follow a normal distribution, the Mann-Whitney U test was applied because of its suitability for comparing two independent groups with nonparametric data. For normally distributed variables, Student's t test was used to compare means between the COVID-19-positive and COVID-19-negative groups. Logistic regression was employed to evaluate the association between waiting time intervals (as a continuous predictor) and postoperative pulmonary complications (a binary outcome), given its robustness for such analyses. Categorical data, such as operation types and comorbidities, were compared via the chi-square test or Fisher's exact test when expected cell counts were low, ensuring statistical validity. A p value <0.05 was considered to indicate statistical significance. Compared with experimental models such as D'Albo et al.[21] (n = 82), which effectively identified significant effects of mechanical power, our sample size of 110 patients was adequate to detect differences in lung dynamics. Patients were monitored with a bispectral index (BIS) (Covidien, Boulder, CO, USA) and Train-of-Four (TOF) (GE HealthCare, Chicago, Illinois, USA) in addition to the monitoring recommended by the American Society of Anesthesiologist (ASA). Patients were given IV access with a 22G branch contralateral to the side to be operated on. After preoxygenation with 80% FiO2, anesthesia was induced with 1 mg/kg lidocaine and 1.5 mcg/kg fentanyl followed by propofol under BIS guidance, and 1.2 mg/kg rocuronium was administered after the reference value for TOF was taken. After TOF 0 was observed, patients were intubated with a double lumen tube with a Macintosh blade. The size of the tube was determined to be 35-37 Fr for women and 39-41 Fr for men. The placement of the tube was confirmed via bronchoscopy. Patients were placed in the lateral decubitus position after fixation. After the position was completed, the placement of the tube was confirmed again via bronchoscopy. The mechanical ventilator settings were determined to be 7 ml/kg according to the ideal weight for both lungs and 5 ml/kg for single-lung ventilation. The PEEP (positive end-expiration pressure) was set as 5 cm H2O for all of the patients. FiO2 was titrated to a SpO2 >92. Mechanical power (MP) was calculated via the simplified formula of Gattinoni et al.: MP = 0.098 × RR × VT × (Ppeak - Pplat/2), where RR is the respiratory rate, VT is the tidal volume, Ppeak is the peak pressure, and Pplat is the plateau pressure. This measures the energy delivered to the lungs during ventilation, expressed in joules/minute.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years and planned procedures, including pneumonectomy, lobectomy, segmentectomy, or other lung resections

Exclusion Criteria:

* patient refusal to participate and inability to provide informed consent due to psychological or mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated for thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Mechanical Power Calculation | Intraoperative period ( Day of Surgery)

SECONDARY OUTCOMES:
Plato Pressure | Intraoperative period ( Day of Surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No